CLINICAL TRIAL: NCT03286153
Title: Comparison of Ideal vs. Actual Weight Base Factor Dosing
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bloodworks (Other)
Collaborators: Seattle Children's Hospital (Other); Oregon Health and Science University (Other); Providence Health & Services (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: BDC Ideal Body Weight Dosing
Record Dates: First submitted 2017-08-09; First posted 2017-09-18 (Actual); Last update posted 2017-09-18 (Actual); Status verified 2017-09

CONDITIONS: Hemophilia A
Keywords: Hemophilia A; FVIII; Ideal body weight; Actual body weight
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Intervention Model Description: Subjects are randomized to receive factor based either on ideal body weight or actual body weight first followed by receiving factor based on the other category next
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ideal Body Weight First (Experimental): Randomized to receive factor product based on ideal body weight first
  Interventions: Other: Ideal Body Weight First
- Actual Body Weight First (Experimental): Randomized to receive factor product based on actual body weight first
  Interventions: Other: Actual Body Weight First

INTERVENTIONS:
Other: Ideal Body Weight First — Randomized to receive 50 U/kg (+/- 20%) of the factor product participants routinely use based on ideal body weight. For participants age 12-19, ideal weight is calculated using the McLaren method. For participants age 20 and over, ideal weight is calculated using the following equation: [50kg + (2.3kg*every inch over 5 feet)].
  Arms: Ideal Body Weight First
Other: Actual Body Weight First — Randomized to receive 50 U/kg (+/- 20%) of the factor product participants routinely use based on actual body weight.
  Arms: Actual Body Weight First

SUMMARY:
This is a randomized, prospective, multicenter study to examine whether or not the current recommended factor dosing strategy - i.e., dosing by actual body weight - in overweight and obese patients with Hemophilia A may deliver excessive clotting factor to achieve the desired result of bleeding prevention and cessation. This study also examines ways to prevent delivering excessive factor by using a patient's ideal body weight as a new dosing strategy compared to the current dosing strategy. The hypothesis being tested is that factor dosing based on ideal body weight will result in protective factor levels.

DETAILED DESCRIPTION:
This is a randomized, prospective, multicenter, open-label, crossover study to examine whether or not the current recommended factor dosing strategy, i.e., dosing by actual body weight in overweight and obese patients, may deliver more clotting factor than necessary to cause bleeding to stop in participants with Hemophilia A who use Factor VIII (FVIII). This study also examines ways to prevent delivering too much factor by using a participant's ideal body weight as a new dosing strategy compared to the current dosing strategy. The hypothesis being tested is that factor dosing based on ideal body weight will result in hemostatic factor levels.

The study will be conducted at the Washington Center for Bleeding Disorders (WCBD) at Bloodworks Northwest, Oregon Health & Science University (OHSU), Seattle Children's Hospital (SCH), and Providence Sacred Heart Children's Hospital (SH). Cumulatively across the four sites, up to 20 participants will be enrolled. Randomization will be performed centrally at WCBD.

Participants will provide their own factor. Prior to the first study-related dose, participants will stop taking any FVIII products for either 48 hours if currently using a short-acting FVIII product or 72 hours for a long acting FVIII product. Factor levels will be measured immediately before and at multiple points after two different factor doses. Subjects will be randomized to start their dosage based either on actual body weight or ideal body weight first and then crossover to receive dosage based on the other category.

ELIGIBILITY:
Inclusion Criteria:

* Hemophilia A
* Able and willing to comply with pharmacokinetic testing schedule
* Either overweight or obese BMI using CDC definitions by age

Exclusion Criteria:

* Inhibitor of > 0.6 BU twice in the past, or documented abnormal recovery of less than 66% (of expected) in the past
* Known other bleeding disorder
* Known other prolongation in aPTT (lupus anticoagulant, FXII deficiency)
* Female

Min Age: 12 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-01 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Recovery | Change from baseline at up to two months
  Compare the recovery with FVIII between doses calculated on actual body weight versus ideal body weight in subjects with Hemophilia A
Underdosing | Change from baseline at up to two months
  Determine the likelihood of underdosing when using ideal body weight
Overdosing | Change from baseline at up to two months
  Determine the likelihood of overdosing when using actual body weight

SECONDARY OUTCOMES:
Effect of half-life | Change from baseline at up to two months
  Determine the effect on half-life of these dosing strategies
Effect on hemophilia severity | Change from baseline at 20-40 minutes, 5-7 hours, 20-26 hours, and 44-50 hours for both half-life and extended half-life and also at 69-75 hours, and 93-99 hours for extended half-life
  Determine the effect of pharmacokinetic differences on hemophilia severity
Regular half-life vs. extended half-life Regular half-life vs. extended half-life | Change from baseline at up to two months
  Determine differences in participants receiving regular half-life versus extended half-life products
Overweight vs. obese | Change from baseline at up to two months
  Determine the differences, if any, between overweight and obese participants

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Kruse-Jarres, MD, MPH, Principal Investigator — Washington Center for Bleeding Disorders at Bloodworks Northwest
Locations (4):
- United States (4):
  - Oregon Health & Science University, Portland, Oregon
  - Washington Center for Bleeding Disorders at Bloodworks Northwest, Seattle, Washington
  - Seattle Children's Hospital, Seattle, Washington
  - Providence Sacred Heart Children's Hospital, Spokane, Washington

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (5):
  • Informed Consent Form: Main (2017-08-07): https://cdn.clinicaltrials.gov/large-docs/53/NCT03286153/ICF_000.pdf
  • Informed Consent Form: Consent/Assent SC (2017-08-07): https://cdn.clinicaltrials.gov/large-docs/53/NCT03286153/ICF_001.pdf
  • Informed Consent Form: Assent Age 15 to 17 (2017-08-07): https://cdn.clinicaltrials.gov/large-docs/53/NCT03286153/ICF_002.pdf
  • Informed Consent Form: Assent Age 7 to 14 (2017-08-07): https://cdn.clinicaltrials.gov/large-docs/53/NCT03286153/ICF_003.pdf
  • Study Protocol (2016-10-12): https://cdn.clinicaltrials.gov/large-docs/53/NCT03286153/Prot_004.pdf